CLINICAL TRIAL: NCT03040817
Title: Cooperative Group for Clinical Research in G-POEM (POP), Jiangsu, China
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Ruihua Shi, MD, PhD, Postdoctoral Mentor, Chief Physician, Zhongda Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GI of ZhongdaH
Record Dates: First submitted 2017-01-31; First posted 2017-02-02 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Gastric Peroral Endoscopic Pyloromyotomy (G-POEM)
MeSH Terms: interventions — Pyloromyotomy; Esomeprazole; mosapride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- G-POEM (Experimental): Each participant receive gastric peroral endoscopic pyloromyotomy (G-POEM).
  Interventions: Procedure: Gastric peroral endoscopic pyloromyotomy (G-POEM)
- Esomeprazole + Mosapride (Active Comparator): Each participant receive Esomeprazole+ Mosapride. The dosages are：Nexium 40mg bid， Mosapride Citrate Tablets 5mg tid.
  Interventions: Drug: Esomeprazole + Mosapride

INTERVENTIONS:
Procedure: Gastric peroral endoscopic pyloromyotomy (G-POEM) — G-POEM procedure:
  A. Premixed methylene blue/normal saline were injected into gastric antrum submucosa at greater curvature, 5 cm proximal to the pylorus.
  B. Submucosal tunnel was created via endoscopic submucosal dissection. C. A white thick pyloric band, was in contrast to a thin-walled submucosal space of the duodenum observed distally.
  D. Pyloromyotomy starts with dissection of the pyloric ring exposing muscular layer underneath.
  E. Circular and longitudinal myotomy for 2-3 cm. F. Serosa indicates appropriate depth of myotomy. G. Reevaluation of the mucosotomy site. H. Mucosal entry was closed with clips from distal mucosal incision point.
  Other Names: Peroral endoscopic pyloromyotomy (POP)
  Arms: G-POEM
Drug: Esomeprazole + Mosapride — Each participant receive Esomeprazole （Nexium） 40mg bid + Mosapride （Mosapride Citrate Tablets） 5mg tid.
  Other Names: Nexium + Mosapride Citrate Tablets
  Arms: Esomeprazole + Mosapride

SUMMARY:
Diabetic gastroparesis, postsurgical gastroparesis, idiopathic gastroparesis and primary pyloric stenosis are debilitating gastrointestinal motility disorder. However, there is limited medical therapeutic options for these diseases. Gastric peroral endoscopic pyloromyotomy (G-POEM) is an emerging novel endoscopic technique which is reported as a minimally invasive therapy. But so far, the efficacy and safety of G-POEM on these diseases are rarely explored. So, there is a cooperative group composed of five clinical centers for clinical research in G-POEM.

DETAILED DESCRIPTION:
Participants are randomly devided into 'G-POEM group' and 'Esomeprazole+Mosapride group'. In G-POEM group, each participant receives G-POEM treatment. In Esomeprazole+Mosapride group, each participant receives Nexium 40mg bid + Mosapride Citrate Tablets 5mg tid. The whole outcome measure time fram is up to two years. Outcome evaluations include: gastric emptying imaging, gastric antrum volume, gastric emptying time, gastroparesis cardinal symptoms index and gastroesophageal reflux disease questionnaire. All the outcomes are assessed at different time points (from baseline to 6 months, 12months and 24months).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 16 to 80 years old
2. Full sufficiency in literacy
3. Be off proton pump inhibitor, antacids and prokinetics ≥ 2 weeks
4. Refractory gastroesophageal reflux disease induced by postsurgical gastroparesis

Exclusion Criteria:

1. Severe heart, lung, and cerebrovascular disease
2. Severe hematopoietic system disease
3. Abnormal blood coagulation function
4. Oropharyngeal abnormalities
5. Severe spine malformation
6. In pregnancy and lactation at present, or plan to become pregnant within 2 years
7. Severe inflammation or huge ulcers in stomach
8. Mental and psychological disorder

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2019-08-16 (Estimated); Study Completion 2019-12-16 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Gastric Emptying Imaging at 6 months. | From baseline to 6 months.
  Each participant will receive gastric emptying imaging measurement both at baseline and 6 months.
Change from Baseline in Gastric Emptying Imaging at 12 months. | From baseline to 12 months.
  Each participant will receive gastric emptying imaging measurement both at baseline and 12 months.
Change from Baseline in Gastric Emptying Imaging at 24 months. | From baseline to 24 months.
  Each participant will receive gastric emptying imaging measurement both at baseline and 24 months.
Change from Baseline in Gastric Antrum Volume at 6 months. | From baseline to 6 months.
  Each participant will receive gastric antrum volume measurement both at baseline and 6 months.
Change from Baseline in Gastric Antrum Volume at 12 months. | From baseline to 12 months.
  Each participant will receive gastric antrum volume measurement both at baseline and 12 months.
Change from Baseline in Gastric Antrum Volume at 24 months. | From baseline to 24 months.
  Each participant will receive gastric antrum volume measurement both at baseline and 24 months.
Change from Baseline in Gastric Emptying Time at 6 months. | From baseline to 6 months.
  Each participant will receive gastric emptying time measurement both at baseline and 6 months.
Change from Baseline in Gastric Emptying Time at 12 months. | From baseline to 12 months.
  Each participant will receive gastric emptying time measurement both at baseline and 12 months.
Change from Baseline in Gastric Emptying Time at 24 months. | From baseline to 24 months.
  Each participant will receive gastric emptying time measurement both at baseline and 24 months.
Change from Baseline in Gastroparesis Cardinal Symptoms Index at 6 months. | From baseline to 6 months.
  Each participant will receive gastroparesis cardinal symptoms index evaluation both at baseline and 6 months.
Change from Baseline in Gastroparesis Cardinal Symptoms Index at 12 months. | From baseline to 12 months.
  Each participant will receive gastroparesis cardinal symptoms index evaluation both at baseline and 12 months.
Change from Baseline in Gastroparesis Cardinal Symptoms Index at 24 months. | From baseline to 24 months.
  Each participant will receive gastroparesis cardinal symptoms index evaluation both at baseline and 24 months.
Change from Baseline in Gastroesophageal Reflux Disease Questionnaire at 6 months. | From baseline to 6 months.
  Each participant will receive gastroesophageal reflux disease questionnaire evaluation both at baseline and 6 months.
Change from Baseline in Gastroesophageal Reflux Disease Questionnaire at 12 months. | From baseline to 12 months.
  Each participant will receive gastroesophageal reflux disease questionnaire evaluation both at baseline and 12 months.
Change from Baseline in Gastroesophageal Reflux Disease Questionnaire at 24 months. | From baseline to 24 months.
  Each participant will receive gastroesophageal reflux disease questionnaire evaluation both at baseline and 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Huiping Wang, Study Chair — Zhongda Hospital
Locations (1):
- Zhongda Hospital Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided